CLINICAL TRIAL: NCT02411448
Title: A Multicenter, Randomized, Double-Blind Study of Erlotinib in Combination With Ramucirumab or Placebo in Previously Untreated Patients With EGFR Mutation-Positive Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Ramucirumab (LY3009806) in Combination With Erlotinib in Previously Untreated Participants With EGFR Mutation-Positive Metastatic NSCLC (RELAY)
Acronym: RELAY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15540; I4T-MC-JVCY (Other: Eli Lilly and Company); 2014-004824-22 (EudraCT Number)
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ramucirumab; Erlotinib Hydrochloride; Gefitinib; osimertinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ramucirumab + Erlotinib (Experimental): Part A: 10 milligrams per kilogram (mg/kg) ramucirumab administered every 2 weeks intravenously (IV) in combination with 150 mg erlotinib daily orally.
  Participants may continue to receive treatment until discontinuation criteria are met.
  Part B: 10 mg/kg ramucirumab administered every 2 weeks IV in combination with 150 mg erlotinib daily orally. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab; Drug: Erlotinib
- Placebo + Erlotinib (Placebo Comparator): Part B: Placebo administered every 2 weeks IV in combination with 150 mg erlotinib daily orally.
  Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Placebo; Drug: Erlotinib
- Ramucirumab + Gefitinib or Osimertinib (Experimental): Part C: 10 mg/kg ramucirumab administered every 2 weeks intravenously (IV) + 250 mg Gefitinib or 80 mg Osimertinib daily orally.
  * Ramucirumab and gefitinib administered during period 1.
  * Ramucirumab and osimertinib administered during period 2.
  Interventions: Drug: Ramucirumab; Drug: Gefitinib; Drug: Osimertinib

INTERVENTIONS:
Drug: Ramucirumab — Administered IV.
  Other Names: LY3009806
  Arms: Ramucirumab + Erlotinib; Ramucirumab + Gefitinib or Osimertinib
Drug: Placebo — Administered IV.
  Arms: Placebo + Erlotinib
Drug: Erlotinib — Administered orally.
  Arms: Placebo + Erlotinib; Ramucirumab + Erlotinib
Drug: Gefitinib — Administered orally.
  Arms: Ramucirumab + Gefitinib or Osimertinib
Drug: Osimertinib — Administered orally.
  Arms: Ramucirumab + Gefitinib or Osimertinib

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of ramucirumab in combination with erlotinib as compared to placebo in combination with erlotinib in previously untreated participants with stage IV non-small cell lung cancer (NSCLC) harboring an activating epidermal growth factor receptor (EGFR) mutation (Exon 19-Del and Exon 21 L858R). Safety and tolerability of ramucirumab in combination with erlotinib will be assessed in Part A before proceeding to Part B.

The purpose of Part C is to determine the efficacy and safety of ramucirumab in combination with gefitinib in previously untreated East Asian participants with EGFR mutation-positive metastatic NSCLC and of ramucirumab in combination with osimertinib in those participants whose disease progressed on ramucirumab and gefitinib and that have T790M - positive metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed diagnosis of Stage IV NSCLC as defined by the American Joint Committee on Cancer Staging Criteria for Lung Cancer (AJCC 7th edition 2009).
* Eligible for first-line treatment with erlotinib based on documented evidence of tumor harboring an activating EGFR mutation [exon 19 deletion or exon 21 (L858R) substitution mutation].
* Mandatory provision of adequate archived stage IV NSCLC tissue samples or tissue samples other than stage IV NSCLC may be acceptable (optional for part C).
* At least one measurable lesion.
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Known T790M EGFR mutation (not applicable for Part C Period 2).
* Known leptomeningeal carcinomatosis, uncontrolled/unstable spinal cord compression, or brain metastases.
* Serious illness or medical condition.
* Ongoing treatment with CYP3A4 inducers or strong inhibitors.
* Ongoing therapy with nonsteroidal anti-inflammatory drugs for more than 2 months.
* History of gross hemoptysis.
* Significant bleeding disorders.
* Radiologically documented evidence of major blood vessel invasion or encasement by cancer.
* Radiographic evidence of intratumor cavitation.
* History of gastrointestinal perforation within last 6 months.
* History of bowel obstruction, inflammatory enteropathy or extensive intestinal resection.
* History of any arterial thrombotic event within 6 months prior to enrollment.
* The participant has any known significant ophthalmologic abnormalities of the surface of the eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (106):
- United States (7):
  - UCLA Hematology/Oncology - Santa Monica, Los Angeles, California
  - St. Charles Health System, Denver, Colorado
  - The Gastroenterology Group, P.C., Honolulu, Hawaii
  - Cancer Center of Kansas, Wichita, Kansas
  - Queens Medical Associates, Fresh Meadows, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - AHN Allegheny General Hospital, Pittsburgh, Pennsylvania
- Cross Cancer Institute, Edmonton, Alberta, Canada
- France (5):
  - Hôpital Arnaud de Villeneuve - CHU Montpellier, Montpellier, Hérault
  - Chu Grenoble Alpes, La Tronche, Isère
  - Hopital Claude Huriez - CHU de Lille, Lille, Nord
  - Centre Hospitalier Universitaire de Poitiers, Poitiers, Vienne
  - Hôpital Européen Georges Pompidou, Paris
- Germany (7):
  - Robert-Bosch-Krankenhaus, Gerlingen, Baden-Wurttemberg
  - Thoraxklinik Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg
  - Klinikum Köln-Merheim, Cologne, North Rhine-Westphalia
  - Klinikum Chemnitz GmbH, Chemnitz, Saxony
  - Städtisches Krankenhaus Martha-Maria Halle-Dölau gGmbH, Halle, Saxony-Anhalt
  - LungenClinic Grosshansdorf, Großhansdorf, Schleswig-Holstein
  - Helios Klinikum Emil von Behring Berlin-Zehlendorf, Berlin
- Sotiria Thoracic Diseases Hospital of Athens, Athens, Attikí, Greece
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Queen Elizabeth Hospital, Yau Ma Tei
- Italy (6):
  - Instituto Tumori Giovanni Paolo II, Bari, Apulia
  - Cro-Irccs, Aviano, Friuli Venezia Giulia
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga, Orbassano, Torino
  - IRCCS - AOU di Bologna, Bologna
  - Ospedale San Raffaele, Milan
  - Istituto Oncologico Veneto IRCCS, Padua
- Japan (41):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Ehime University Hospital, Tōon, Ehime
  - Kurume University Hospital, Kurume, Fukuoka
  - National Hospital Organization Asahikawa Medical Center, Asahikawa, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Hyogo Prefectual Amagasaki General Medical Center, Amagashiki, Hyōgo
  - Himeji Medical Center, Himeji, Hyōgo
  - Foundation for Biomedical Research and innovation, Kobe, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Osaka Habikino Medical Center, Habikino, Osaka
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Kishiwada City Hospital, Kishiwada, Osaka
  - Kindai University Hospital- Osakasayama Campus, Ōsaka-sayama, Osaka
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai, Osaka
  - Saitama Prefectural Cancer Center, Ina-machi, Saitama
  - Shizuoka Cancer Center, Nakatogari, Shizuoka
  - Tokyo Met Cancer & Infectious Diseases Center Komagome Hp, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - National Hospital Organization Yamaguchi Ube Medical Center, Ube, Yamaguchi
  - Chiba University Hospital, Chiba
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Kyoto University Hospital, Kyoto
  - Nagasaki University Hospital, Nagasaki
  - Niigata University Medical & Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Osaka City General Hospital, Osaka
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka
  - Osaka City University Hospital, Osaka
  - St. Lukes International Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Wakayama MedicaL University Hospital, Wakayama
- Romania (2):
  - Institutul Oncologic, Bucharest, București
  - S.C. MedisProf SRL, Cluj-Napoca, Cluj
- South Korea (10):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbuk-do [Chungbuk]
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - The Catholic University Of Korea St. Vincent's Hospital, Suwon, Kyǒnggi-do
  - Ajou University Hospital, Suwon, Kyǒnggi-do
  - Gyeongsang National University Hospital, Jinju, Kyǒngsangnam-do
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Korea University Guro Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Ulsan University Hospital, Ulsan, Ulsan-Kwangyǒkshi
- Spain (9):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals, Hospitalet, Barcelona [Barcelona]
  - Hospital Son Llatzer, Palma, Illes Balears [Islas Baleares]
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Clinica Universitaria De Navarra, Pamplona, Navarre
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (8):
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - E-DA Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - MacKay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (4):
  - Ege Universitesi Hastanesi, Bornova, İzmir
  - Baskent University Dr. Turgut Noyan Research and Training Center, Adana
  - Trakya University, Edirne
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi Eğitim ve Araştırma Hastanesi, Malatya
- United Kingdom (3):
  - Royal Marsden Hospital (Chelsea), London, Kensington and Chelsea
  - Charing Cross Hospital, Chelsea, London
  - City Hospital, Nottingham University Hospitals, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Nishino K, Seto T, Nishio M, Nishio K, Kasahara K, Satouchi M, Yoh K, Hayashi H, Enatsu S, Matsui T, Varughese SC, Visseren-Grul C, Nakagawa K. RELAY: safety and efficacy of ramucirumab plus erlotinib in elderly Japanese patients with metastatic EGFR-mutated NSCLC. Future Oncol. 2025 Oct;21(24):3197-3206. doi: 10.1080/14796694.2025.2560225. Epub 2025 Sep 25. PMID 40995949
- [Derived] Nishio M, Seto T, Reck M, Garon EB, Nishio K, Kasahara K, Nishino K, Satouchi M, Yoh K, Hayashi H, Sakai K, Enatsu S, Frimodt-Moller B, Matsui T, Varughese SC, Carlsen M, Visseren-Grul C, Nakagawa K. Final Survival Outcomes With Ramucirumab Plus Erlotinib Versus Placebo Plus Erlotinib in Patients With Untreated EGFR-Mutated Metastatic NSCLC: RELAY Japanese Subset. JTO Clin Res Rep. 2025 Feb 28;6(6):100819. doi: 10.1016/j.jtocrr.2025.100819. eCollection 2025 Jun. PMID 40458541
- [Derived] Nakagawa K, Garon EB, Seto T, Nishio M, Aix SP, Paz-Ares L, Chiu CH, Park K, Novello S, Nadal E, Nishino K, Yoh K, Shih JY, Chik JYK, Moro-Sibilot D, Puri T, Chacko Varughese S, Frimodt-Moller B, Visseren-Grul C, Reck M. RELAY: Final Overall Survival for Erlotinib Plus Ramucirumab or Placebo in Untreated, EGFR-Mutated Metastatic NSCLC. J Thorac Oncol. 2025 Apr;20(4):487-499. doi: 10.1016/j.jtho.2024.11.032. Epub 2024 Nov 30. PMID 39622410
- [Derived] Nishio K, Sakai K, Nishio M, Seto T, Visseren-Grul C, Carlsen M, Matsui T, Enatsu S, Nakagawa K. Impact of ramucirumab plus erlotinib on circulating cell-free DNA from patients with untreated metastatic non-small cell lung cancer with EGFR-activating mutations (RELAY phase 3 randomized study). Transl Lung Cancer Res. 2023 Aug 30;12(8):1702-1716. doi: 10.21037/tlcr-22-736. Epub 2023 Aug 10. PMID 37691865
- [Derived] Garon EB, Reck M, Nishio K, Heymach JV, Nishio M, Novello S, Paz-Ares L, Popat S, Aix SP, Graham H, Butts BD, Visseren-Grul C, Nakagawa K; RELAY study investigators. Ramucirumab plus erlotinib versus placebo plus erlotinib in previously untreated EGFR-mutated metastatic non-small-cell lung cancer (RELAY): exploratory analysis of next-generation sequencing results. ESMO Open. 2023 Aug;8(4):101580. doi: 10.1016/j.esmoop.2023.101580. Epub 2023 Jun 28. PMID 37390764
- [Derived] Chiu CH, Lin MC, Wei YF, Chang GC, Su WC, Hsia TC, Su J, Wang AK, Jen MH, Puri T, Shih JY. Efficacy and Tolerability of Ramucirumab Plus Erlotinib in Taiwanese Patients with Untreated, Epidermal Growth Factor Receptor-Mutated, Stage IV Non-small Cell Lung Cancer in the RELAY Study. Target Oncol. 2023 Jul;18(4):505-515. doi: 10.1007/s11523-023-00975-5. Epub 2023 Jun 17. PMID 37329423
- [Derived] Nakagawa K, Garon EB, Gao L, Callies S, Zimmermann A, Walgren R, Visseren-Grul C, Reck M. RELAY, ramucirumab plus erlotinib versus placebo plus erlotinib in untreated EGFR-mutated metastatic non-small cell lung cancer: exposure-response relationship. Cancer Chemother Pharmacol. 2022 Aug;90(2):137-148. doi: 10.1007/s00280-022-04447-x. Epub 2022 Jul 16. PMID 35841410
- [Derived] Nishio M, Nishio K, Reck M, Garon EB, Imamura F, Kawaguchi T, Yamaguchi H, Ikeda S, Hirano K, Visseren-Grul C, Ceccarelli M, Wijayawardana SR, Zimmermann A, Matsui T, Enatsu S, Nakagawa K. RELAY+: Exploratory Study of Ramucirumab Plus Gefitinib in Untreated Patients With EGFR-Mutated Metastatic NSCLC. JTO Clin Res Rep. 2022 Feb 26;3(4):100303. doi: 10.1016/j.jtocrr.2022.100303. eCollection 2022 Apr. PMID 35369607
- [Derived] Nadal E, Horinouchi H, Shih JY, Nakagawa K, Reck M, Garon EB, Wei YF, Kollmeier J, Frimodt-Moller B, Barrett E, Lipkovich O, Visseren-Grul C, Novello S. RELAY, Ramucirumab Plus Erlotinib Versus Placebo Plus Erlotinib in Patients with Untreated, Epidermal Growth Factor Receptor Mutation-Positive, Metastatic Non-Small-Cell Lung Cancer: Safety Profile and Manageability. Drug Saf. 2022 Jan;45(1):45-64. doi: 10.1007/s40264-021-01127-2. Epub 2021 Dec 20. PMID 34928484
- [Derived] Mitani S, Chen Y, Inoue K, Mori J, Gao L, Long A, Wakabayashi S. Clinical Impact of a Shortened Infusion Duration of Ramucirumab in Japanese Patients -A Model-Based Approach. Gan To Kagaku Ryoho. 2021 Nov;48(11):1381-1387. PMID 34795131
- [Derived] Nakagawa K, Garon EB, Seto T, Nishio M, Ponce Aix S, Paz-Ares L, Chiu CH, Park K, Novello S, Nadal E, Imamura F, Yoh K, Shih JY, Au KH, Moro-Sibilot D, Enatsu S, Zimmermann A, Frimodt-Moller B, Visseren-Grul C, Reck M; RELAY Study Investigators. Ramucirumab plus erlotinib in patients with untreated, EGFR-mutated, advanced non-small-cell lung cancer (RELAY): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2019 Dec;20(12):1655-1669. doi: 10.1016/S1470-2045(19)30634-5. Epub 2019 Oct 4. PMID 31591063
- [Derived] Reck M, Garon EB, Paz-Ares L, Ponce S, Jaime JC, Juan O, Nadal E, Kiura K, Widau RC, He S, Dalal R, Lee P, Nakagawa K. Randomized, Double-Blind Phase Ib/III Study of Erlotinib With Ramucirumab or Placebo in Previously Untreated EGFR-Mutant Metastatic Non-Small-Cell Lung Cancer (RELAY): Phase Ib Results. Clin Lung Cancer. 2018 May;19(3):213-220.e4. doi: 10.1016/j.cllc.2017.11.003. Epub 2017 Nov 21. PMID 29317191
- [Derived] Garon EB, Reck M, Paz-Ares L, Ponce S, Jaime JC, Juan O, Nadal E, Lee P, Dalal R, Liu J, He S, Treat J, Nakagawa K. Treatment Rationale and Study Design for the RELAY Study: A Multicenter, Randomized, Double-Blind Study of Erlotinib With Ramucirumab or Placebo in Patients With Epidermal Growth Factor Receptor Mutation-Positive Metastatic Non-Small-Cell Lung Cancer. Clin Lung Cancer. 2017 Jan;18(1):96-99. doi: 10.1016/j.cllc.2016.05.023. Epub 2016 Jun 8. PMID 27894601
- See also: A Study of Ramucirumab (LY3009806) in Combination With Erlotinib in Participants With EGFR Mutation-Positive Metastatic NSCLC — https://trials.lillytrialguide.com/en-US/trial/3pxvd64nCo8AmAgMMu6iSo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consists of 3 parts:
  * Part A: Open-label.
  * Part B: Randomized, double-blind and placebo-controlled.
  * Part C: Open-label.
  Part C data will be reported after study completion.
Groups:
- Part A: Ramucirumab + Erlotinib: Part A: 10 milligrams per kilogram (mg/kg) ramucirumab administered every 2 weeks intravenously (IV) in combination with 150 mg erlotinib daily orally.
  Participants may continue to receive treatment until discontinuation criteria are met.
- Part B: Ramucirumab+ Erlotinib: Part B: 10 mg/kg ramucirumab administered every 2 weeks IV in combination with 150 mg erlotinib daily orally.
  Participants may continue to receive treatment until discontinuation criteria are met.
- Part B: Placebo+ Erlotinib: Part B: Placebo administered every 2 weeks IV in combination with 150 mg erlotinib daily orally.
  Participants may continue to receive treatment until discontinuation criteria are met.
Period: Overall Study
Arm/Group | Part A: Ramucirumab + Erlotinib | Part B: Ramucirumab+ Erlotinib | Part B: Placebo+ Erlotinib
Started | 14 | 224 | 225
Received at Least One Dose of Study Drug | 14 | 221 | 225
Completed | 10 | 141 | 173
Not Completed | 4 | 83 | 52
Not completed — Withdrawal by Subject | 1 | 14 | 9
Not completed — Other | 0 | 2 | 0
Not completed — Did not receive study treatment | 0 | 3 | 0
Not completed — Alive on study treatment | 3 | 64 | 43

BASELINE CHARACTERISTICS:
Population: All enrolled participants. Part C data will be reported after study completion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Ramucirumab + Erlotinib | Part B: Ramucirumab+ Erlotinib | Part B: Placebo+ Erlotinib | Total
Number analyzed (Participants) | 14 | 224 | 225 | 463
Age, Continuous [Mean (Standard Deviation); unit: years]
  Part A | 67.6 (13.2) | NA (NA) — Row represents Part A data only. | NA (NA) — Row represents Part A data only. | 67.6 (13)
  Part B | NA (NA) — Row represents Part B data only. | 63.7 (10.2) | 62.9 (10.6) | 63.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 141 | 142 | 294
  Male | 3 | 83 | 83 | 169
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 13 | 10 | 23
  Not Hispanic or Latino | 1 | 150 | 160 | 311
  Unknown or Not Reported | 13 | 61 | 55 | 129
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 7 | 172 | 174 | 353
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 7 | 52 | 48 | 107
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 0 | 2 | 0 | 2
  Hong Kong | 0 | 9 | 6 | 15
  United States | 0 | 7 | 2 | 9
  Japan | 7 | 106 | 105 | 218
  United Kingdom | 0 | 4 | 3 | 7
  Spain | 7 | 23 | 19 | 49
  Canada | 0 | 0 | 2 | 2
  South Korea | 0 | 25 | 29 | 54
  Turkey | 0 | 3 | 4 | 7
  Taiwan | 0 | 26 | 30 | 56
  Italy | 0 | 8 | 12 | 20
  France | 0 | 4 | 7 | 11
  Germany | 0 | 7 | 6 | 13
Geographic Region [Count of Participants; unit: Participants] — * Geographic region "Other" includes Canada, France, Germany, Italy, Romania, Spain, Turkey, US, UK.
  Participants
    East Asia | 7 | 166 | 170 | 343
    Other* | 7 | 58 | 55 | 120

OUTCOME MEASURES:

1. Primary Outcome: Part B: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization to the date of radiographically documented progressive disease (PD) based on investigator assessment, or the date of death due to any cause, whichever is first assessed via Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1 or more new lesions is also considered progression.
Time Frame: Randomization to Measured Progressive Disease or Death from Any Cause (Up To 37 Months)
Population: Part B: All randomized participants grouped according to their assigned treatment at randomization. Censored participants were: Part B: Ramucirumab+ Erlotinib= 102 and Part B: Placebo+ Erlotinib= 67. Per protocol, Part A did not evaluate efficacy.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Ramucirumab+ Erlotinib | Part B: Placebo+ Erlotinib
Number analyzed (Participants) | 224 | 225
Months | 19.4 [15.4 to 21.6] | 12.4 [11.0 to 13.5]
Statistical Analysis 1: Comparison: Part B: Ramucirumab+ Erlotinib vs Part B: Placebo+ Erlotinib; Test type: Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.591, 95% CI 2-sided [0.461 to 0.760]

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section.
Time Frame: Cycle 1 Day 1 through End of Study (Up To 3 Years)
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Ramucirumab + Erlotinib: Part B: 10 mg/kg ramucirumab administered every 2 weeks IV in combination with 150 mg erlotinib daily orally.
  Participants may continue to receive treatment until discontinuation criteria are met.
- Part B: Placebo + Erlotinib: Part B: Placebo administered every 2 weeks IV in combination with 150 mg erlotinib daily orally.
  Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part A: Ramucirumab + Erlotinib | Part B: Ramucirumab + Erlotinib | Part B: Placebo + Erlotinib
Number analyzed (Participants) | 14 | 221 | 225
Participants | 14 | 221 | 225

3. Secondary Outcome: Part B: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. For each participant who was not known to have died as of the data-inclusion cutoff date for a particular analysis,OS was censored for that analysis at the date of last contact prior to the data-inclusion cutoff date (contacts considered in the determination of last contact date include adverse event (AE) date, lesion assessment date, visit date, and last known alive date).
Time Frame: Randomization to Date of Death from Any Cause (Up To 37 Months)
Population: Part B: All randomized participants grouped according to their assigned treatment at randomization. Censored participants were: Part B: Ramucirumab+ Erlotinib= 187 and Part B: Placebo+ Erlotinib= 183. Per protocol, Part A did not evaluate efficacy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B: Ramucirumab+ Erlotinib | Part B: Placebo+ Erlotinib
Number analyzed (Participants) | 224 | 225
months | NA [NA to NA] — There were not enough events/deaths to compute a median or 95% confidence interval. | NA [NA to NA] — There were not enough events/deaths to compute a median or 95% confidence interval.
Statistical Analysis 1: Comparison: Part B: Ramucirumab+ Erlotinib vs Part B: Placebo+ Erlotinib; Test type: Other; p = 0.4209, Log Rank; Hazard Ratio (HR) = 0.832, 95% CI 2-sided [0.532 to 1.303]

4. Secondary Outcome: Part B: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Objective Response Rate [ORR])
Description: ORR was defined as the percentage of randomized participants achieving a best overall response of partial response (PR) or complete response (CR) assessed via Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR was defined as the disappearance of all lesions, pathological lymph node reduction in short axis to <10 mm, and normalization of tumor marker levels of non-target lesions. PR was at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1 or more new lesions is also considered progression.
Time Frame: Randomization to Progressive Disease (Up To 37 Months)
Population: Part B: All randomized participants grouped according to their assigned treatment at randomization. Per protocol, Part A did not evaluate efficacy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: Ramucirumab+ Erlotinib | Part B: Placebo+ Erlotinib
Number analyzed (Participants) | 224 | 225
percentage of participants | 76.3 [70.8 to 81.9] | 74.7 [69.0 to 80.3]
Statistical Analysis 1: Comparison: Part B: Ramucirumab+ Erlotinib vs Part B: Placebo+ Erlotinib; Test type: Other; p = 0.7413, Cochran-Mantel-Haenszel

5. Secondary Outcome: Part B: Percentage of Participants With CR, PR, or Stable Disease (SD) (Disease Control Rate [DCR])
Description: DCR was defined as the percentage of randomized participants achieving a best overall response of CR,PR, or stable disease(SD) assessed via Response Evaluation Criteria in Solid Tumors(RECIST) version 1.1. CR was defined as the disappearance of all lesions,pathological lymph node reduction in short axis to <10 mm, and normalization of tumor marker levels of non-target lesions.PR was at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters.SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease(PD) was at least a 20% increase in the sum of the diameters of target lesions,taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.The appearance of 1 or more new lesions is also considered progression.
Time Frame: Randomization to Progressive Disease (Up To 37 Months)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: Ramucirumab+ Erlotinib | Part B: Placebo+ Erlotinib
Number analyzed (Participants) | 224 | 225
percentage of participants | 95.1 [92.3 to 97.9] | 95.6 [92.9 to 98.2]
Statistical Analysis 1: Comparison: Part B: Ramucirumab+ Erlotinib vs Part B: Placebo+ Erlotinib; Test type: Other; p = 1.0000, Cochran-Mantel-Haenszel

6. Secondary Outcome: Part B: Duration of Response (DoR)
Description: DoR was defined as the date of first documented CR or PR (responder) to the date of progressive disease or the date of death due to any cause, whichever was earlier. If a responder was not known to have died or have progressive disease, then the participant was censored at the date of last evaluable tumor assessment.CR was defined as the disappearance of all lesions, pathological lymph node reduction in short axis to <10 mm, and normalization of tumor marker levels of non-target lesions. PR was at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1 or more new lesions is also considered progression.
Time Frame: Date of Complete Response (CR) or Partial Response (PR) to Date of Objective Disease Progression or Death Due to Any Cause (Up To 37 Months)
Population: Part B: All randomized participants grouped according to their assigned treatment at randomization that had a response (CR or PR). Per protocol, Part A did not evaluate efficacy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B: Ramucirumab+ Erlotinib | Part B: Placebo+ Erlotinib
Number analyzed (Participants) | 171 | 168
months | 18.0 [13.9 to 19.8] | 11.1 [9.7 to 12.3]
Statistical Analysis 1: Comparison: Part B: Ramucirumab+ Erlotinib vs Part B: Placebo+ Erlotinib; Test type: Other; p = 0.0003, Log Rank; Hazard Ratio (HR) = 0.619, 95% CI 2-sided [0.477 to 0.805]

7. Secondary Outcome: Part B: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Ramucirumab
Description: Part B: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Ramucirumab
Time Frame: Cycle 2 Day 1: Predose; Cycle 4 Day 1: Predose; Cycle 7 Day 1: Predose; Cycle 14 Day 1
Population: Part B participants who received at least one dose of Ramucirumab+ Erlotinib who had evaluable PK data. Per protocol, Part A did not evaluate PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Groups:
- Part B: Ramucirumab+ Erlotinib: Part B: 10 mg/kg ramucirumab every 2 weeks IV in combination with 150 mg erlotinib daily orally.
  Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part B: Ramucirumab+ Erlotinib
Number analyzed (Participants) | 185
microgram per milliliter (µg/mL)
  Cycle 2 | 39.6 (32)
  Cycle 4: number analyzed (Participants) | 145
  Cycle 4 | 68.5 (37)
  Cycle 7: number analyzed (Participants) | 110
  Cycle 7 | 85.7 (32)
  Cycle 14: number analyzed (Participants) | 59
  Cycle 14 | 99.4 (31)

8. Secondary Outcome: Part B: Number of Participants With Anti-Ramucirumab Antibodies
Description: Part B: Number of Participants With Anti-Ramucirumab Antibodies.
Time Frame: Cycle 1 Predose through Follow-up (Up To 37 Months)
Population: All participants who received at least one dose of study drug. Per protocol, Part A did not evaluate Anti-Ramucirumab Antibodies .
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Ramucirumab+ Erlotinib | Part B: Placebo+ Erlotinib
Number analyzed (Participants) | 221 | 225
Participants | 14 | 18

9. Secondary Outcome: Part B: Best Change From Baseline on the Lung Cancer Symptom Scale (LCSS)
Description: The LCSS consisted of 9 items: 6 items focused on lung cancer symptoms [loss of appetite, fatigue, cough, dyspnea (shortness of breath), hemoptysis (blood in sputum), and pain] and 3 global items (symptom distress, interference with activity level, and global quality of life). Participant responses to each item were measured using visual analogue scales (VAS) with 100-millimeter (mm) lines. A higher score for any item represented a higher level of symptoms/problems. The LCSS total score was defined as the mean of all 9 items. Average symptom burden index (ASBI) was calculated as the mean of the six symptom-specific questions from the LCSS. Potential scores range from 0 (for best outcome) to 100 (for worst outcome).
Time Frame: Baseline, End of Study (Up To 37 Months)
Population: Part B: All randomized participants who completed the LCSS at baseline and at least once post-baseline. Per protocol, Part A did not evaluate efficacy.
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | Part B: Ramucirumab+ Erlotinib | Part B: Placebo+ Erlotinib
Number analyzed (Participants) | 224 | 225
millimeter
  Loss of Appetite: number analyzed (Participants) | 213 | 217
  Loss of Appetite | -17.07 (0.92) | -18.16 (0.91)
  Fatigue: number analyzed (Participants) | 213 | 217
  Fatigue | -19.35 (0.91) | -19.45 (0.90)
  Cough: number analyzed (Participants) | 213 | 217
  Cough | -21.22 (0.58) | -22.09 (0.57)
  Shortness of Breath: number analyzed (Participants) | 213 | 217
  Shortness of Breath | -14.46 (0.57) | -15.93 (0.57)
  Blood in Sputum: number analyzed (Participants) | 213 | 216
  Blood in Sputum | -1.58 (0.25) | -1.94 (0.25)
  Pain: number analyzed (Participants) | 213 | 216
  Pain | -13.57 (0.59) | -14.69 (0.59)
  Symptom distress: number analyzed (Participants) | 213 | 217
  Symptom distress | -15.91 (0.67) | -16.15 (0.67)
  Interference with Activity Level: number analyzed (Participants) | 213 | 217
  Interference with Activity Level | -14.43 (0.83) | -15.60 (0.82)
  Global Quality of Life: number analyzed (Participants) | 213 | 217
  Global Quality of Life | -16.21 (0.95) | -18.12 (0.94)
  Average Symptom Burden Index: number analyzed (Participants) | 213 | 216
  Average Symptom Burden Index | -12.17 (0.57) | -13.05 (0.57)
  Total LCSS: number analyzed (Participants) | 213 | 216
  Total LCSS | -12.00 (0.62) | -12.71 (0.61)

10. Secondary Outcome: Part B: Change From Baseline on the EuroQol 5-Dimension, 5-Level Questionnaire (EQ-5D-5L) Index Score
Description: The EQ-5D-5L is a standardized instrument used to measure self-reported health status of the participants. It consists of 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). There are 5 response levels (no problems, slight problems, moderate problems, severe problems, and extreme problems/unable to), ranging from 1 to 5 (good to bad). Dimension responses were converted to an index score using UK weights. The index scores were anchored on full health (1.0) to dead (0) with negative values assigned to health states considered worse than death.
Time Frame: Baseline, Cycle 10 (each cycle is 2 weeks)
Population: Part B: All randomized participants who completed the EQ-5D-5L at baseline and at least once post-baseline. Per protocol, Part A did not evaluate efficacy.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part B: Placebo+ Erlotinib: Part B: Placebo every 2 weeks IV in combination with 150 mg erlotinib daily orally.
  Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part B: Ramucirumab+ Erlotinib | Part B: Placebo+ Erlotinib
Number analyzed (Participants) | 170 | 170
score on a scale | 0.02 (0.15) | 0.02 (0.15)

11. Secondary Outcome: Part B: Change From Baseline on the EuroQol 5-Dimension, 5-Level Questionnaire (EQ-5D-5L) Index Score
Description: as for outcome 10
Time Frame: Baseline, Cycle 28 (each cycle is 2 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Ramucirumab+ Erlotinib | Part B: Placebo+ Erlotinib
Number analyzed (Participants) | 108 | 81
score on a scale | 0.02 (0.18) | 0.01 (0.1)

12. Secondary Outcome: Part B: Change From Baseline on the EuroQol 5-Dimension, 5-Level Questionnaire (EQ-5D-5L) Index Score
Description: as for outcome 10
Time Frame: Baseline, Cycle 40 (each cycle is 2 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Ramucirumab+ Erlotinib | Part B: Placebo+ Erlotinib
Number analyzed (Participants) | 57 | 44
score on a scale | 0.01 (0.15) | -0.01 (0.14)

ADVERSE EVENTS:
Time Frame: Up To 3 Years
Description: Serious Adverse Events and Other Adverse Events: All participants who received at least one dose of study drug; All-Cause Mortality: All randomized participants. Part C data will be reported after study completion. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | Part A: Ramucirumab + Erlotinib | Part B: Ramucirumab + Erlotinib | Part B: Placebo + Erlotinib
All-Cause Mortality (participants affected / at risk) | 2/14 | 37/224 | 42/225
Serious Adverse Events (participants affected / at risk) | 0/14 | 65/221 | 47/225
Other Adverse Events (participants affected / at risk) | 14/14 | 220/221 | 225/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A: Ramucirumab + Erlotinib (N=14) | Part B: Ramucirumab + Erlotinib (N=221) | Part B: Placebo + Erlotinib (N=225)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Wolff-parkinson-white syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 2 (3)
Macular fibrosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucous membrane disorder (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 4 (4)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 3 (5) | 2 (3)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 4 (5) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Encephalitis influenzal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 7 (9) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (8) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Mesenteric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/11 (0) | 1/139 (1) | 0/142 (0)
Pericarditis malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0/11 (0) | 0/139 (0) | 1/142 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A: Ramucirumab + Erlotinib (N=14) | Part B: Ramucirumab + Erlotinib (N=221) | Part B: Placebo + Erlotinib (N=225)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 21 (49) | 10 (15)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 3 (9) | 2 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (6) | 5 (9) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 2 (3) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 12 (16) | 4 (5)
Hypothyroidism (Endocrine disorders) | 1 (1) | 3 (3) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 4 (7) | 9 (11)
Dry eye (Eye disorders) | 1 (1) | 22 (27) | 23 (24)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 1 (2) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 3 (3) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 15 (26) | 15 (18)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 17 (23) | 19 (41)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 2 (5) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 7 (8) | 5 (5)
Constipation (Gastrointestinal disorders) | 2 (3) | 42 (52) | 31 (38)
Dental caries (Gastrointestinal disorders) | 1 (1) | 8 (8) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 13 (57) | 154 (410) | 160 (388)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 8 (8) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 11 (17) | 12 (21)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 4 (6) | 5 (6)
Gastritis (Gastrointestinal disorders) | 0 (0) | 19 (22) | 9 (11)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 16 (22) | 9 (12)
Gingival bleeding (Gastrointestinal disorders) | 2 (2) | 19 (23) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 14 (19) | 9 (12)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 57 (81) | 44 (79)
Oesophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 6 (13) | 92 (148) | 82 (144)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 5 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (6) | 26 (34) | 25 (31)
Asthenia (General disorders) | 3 (11) | 17 (34) | 14 (29)
Chest pain (General disorders) | 2 (2) | 5 (5) | 3 (3)
Cyst (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (10) | 25 (55) | 27 (51)
Influenza like illness (General disorders) | 0 (0) | 5 (8) | 13 (17)
Malaise (General disorders) | 0 (0) | 34 (69) | 19 (35)
Mucosal inflammation (General disorders) | 2 (3) | 14 (28) | 6 (6)
Non-cardiac chest pain (General disorders) | 1 (1) | 10 (13) | 5 (5)
Oedema (General disorders) | 2 (2) | 3 (4) | 2 (2)
Oedema peripheral (General disorders) | 5 (6) | 50 (78) | 10 (11)
Pain (General disorders) | 1 (1) | 6 (6) | 9 (10)
Pyrexia (General disorders) | 3 (4) | 45 (57) | 24 (34)
Xerosis (General disorders) | 1 (1) | 7 (9) | 4 (5)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 2 (6) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 2 (2)
Angular cheilitis (Infections and infestations) | 1 (1) | 3 (3) | 6 (7)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (6) | 21 (26) | 32 (40)
Cystitis (Infections and infestations) | 1 (1) | 8 (12) | 9 (17)
Eye infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 7 (17) | 11 (15)
Gastroenteritis (Infections and infestations) | 1 (1) | 5 (5) | 4 (4)
Gingivitis (Infections and infestations) | 1 (1) | 6 (16) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (6) | 22 (27) | 18 (28)
Paronychia (Infections and infestations) | 10 (24) | 118 (277) | 114 (238)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Perichondritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 15 (20) | 6 (7)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 6 (12) | 14 (34)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 4 (4) | 4 (4)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 2 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (5) | 38 (53) | 34 (52)
Urinary tract infection (Infections and infestations) | 2 (3) | 17 (23) | 11 (21)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 6 (6)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 7 (12) | 93 (270) | 70 (192)
Aspartate aminotransferase increased (Investigations) | 5 (7) | 92 (270) | 58 (128)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 23 (39) | 20 (46)
Blood bilirubin increased (Investigations) | 3 (4) | 68 (254) | 70 (251)
Blood creatinine increased (Investigations) | 1 (1) | 5 (13) | 6 (8)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 6 (22) | 2 (11)
Electrocardiogram qt prolonged (Investigations) | 1 (2) | 3 (6) | 4 (5)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 12 (35) | 7 (11)
Neutrophil count decreased (Investigations) | 1 (1) | 25 (83) | 16 (39)
Platelet count decreased (Investigations) | 3 (5) | 31 (54) | 6 (10)
Transaminases increased (Investigations) | 1 (1) | 2 (5) | 1 (1)
Weight decreased (Investigations) | 1 (2) | 28 (54) | 29 (37)
White blood cell count decreased (Investigations) | 0 (0) | 14 (53) | 7 (14)
Decreased appetite (Metabolism and nutrition disorders) | 4 (11) | 57 (101) | 47 (84)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 14 (27) | 10 (17)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 18 (38) | 5 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (9) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 24 (28) | 17 (22)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (12) | 8 (11)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (8) | 12 (15)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 12 (14) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (10) | 9 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (8) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 9 (9) | 12 (16)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 4 (5)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (6) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 20 (27) | 19 (24)
Dysgeusia (Nervous system disorders) | 3 (3) | 39 (46) | 32 (44)
Headache (Nervous system disorders) | 7 (13) | 33 (56) | 16 (21)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (3) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 7 (7) | 9 (10)
Anxiety (Psychiatric disorders) | 1 (1) | 7 (16) | 4 (5)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (3) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (2) | 2 (2) | 4 (5)
Insomnia (Psychiatric disorders) | 3 (3) | 32 (36) | 29 (33)
Haematuria (Renal and urinary disorders) | 1 (2) | 10 (11) | 8 (12)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 5 (18) | 75 (278) | 19 (35)
Genital rash (Reproductive system and breast disorders) | 1 (2) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (10) | 48 (62) | 35 (49)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 14 (17) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 18 (25) | 9 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 74 (102) | 27 (33)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 11 (19) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 4 (5) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 19 (25) | 13 (14)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 15 (21) | 11 (17)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 13 (17) | 9 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (7) | 75 (84) | 44 (47)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 9 (33) | 149 (433) | 153 (447)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 6 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (19) | 83 (127) | 91 (181)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 12 (83) | 10 (24)
Hair disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 1/11 (1) | 1/139 (1) | 4/142 (4)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Nail toxicity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (12) | 51 (110) | 66 (165)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2) | 11 (17) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 5 (29) | 39 (103) | 54 (148)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (13) | 20 (47) | 21 (53)
Skin fissures (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (13) | 14 (19)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (4) | 2 (4)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dental care (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Dental operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 2 (3) | 3 (3)
Vaginal pessary insertion (Surgical and medical procedures) | 1/11 (1) | 0/139 (0) | 0/142 (0)
Hypertension (Vascular disorders) | 7 (27) | 100 (246) | 27 (72)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Varicose ulceration (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol: Protocol I4T-MC-JVCY(f) (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT02411448/Prot_000.pdf
  • Study Protocol: Protocol Addendum I4T-MC-JVCY(9) (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT02411448/Prot_002.pdf
  • Statistical Analysis Plan (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT02411448/SAP_001.pdf